CLINICAL TRIAL: NCT06307717
Title: Volatile Anaesthetics on Incidence of Postoperative Depression and Anxiety
Brief Title: Effects of Volatile Anaesthetics on Incidence of Postoperative Depression and Anxiety in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tsinghua Changgeng Hospital (Other); Peking University First Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Xiangya Hospital of Central South University (Other); Beijing Anzhen Hospital (Other); Central South University (Other); Peking University People's Hospital (Other); Zhejiang University (Other); Fudan University (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); China-Japan Friendship Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Taihe Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-DA-002
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Cohort Studies
Keywords: Anxiety; Depression; Aged; Surgery; Volatile anaesthetics
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Sevoflurane; Isoflurane; Desflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- volatile anaesthetic (sevoflurane, isoflurane, desflurane）: Patients receiving volatile anaesthetics received at least one volatile anaesthetic (sevoflurane, isoflurane, desflurane), and those who received non-volatile anaesthetics did not receive any volatile anaesthetic.
  Interventions: Drug: volatile anaesthetic (sevoflurane, isoflurane, desflurane)
- control: Patients receiving volatile anaesthetics received at least one volatile anaesthetic (sevoflurane, isoflurane, desflurane), and those who received non-volatile anaesthetics did not receive any volatile anaesthetic.

INTERVENTIONS:
Drug: volatile anaesthetic (sevoflurane, isoflurane, desflurane) — Patients receiving volatile anaesthetics received at least one volatile anaesthetic (sevoflurane, isoflurane, desflurane), and those who received non-volatile anaesthetics did not receive any volatile anaesthetic.
  Other Names: The blank group was without the use of any inhalation anesthetics
  Groups: volatile anaesthetic (sevoflurane, isoflurane, desflurane）

SUMMARY:
This study is a retrospective analysis of a large-scale multicentre prospective cohort study that investigates the impact of volatile anaesthetics on the incidence of postoperative depression and anxiety among elderly patients.

DETAILED DESCRIPTION:
Studies have suggested volatile anaesthetics may alleviate depression and anxiety in patients. However, there is a paucity of research in this area. The investigatorswanted to determine the association between volatile anaesthetics and depression/anxiety in elderly patients within 7 days after surgery.

This study retrospectively analysed data from a prospective database of patients aged 65 and above who underwent non-cardiac, non-neurosurgical elective surgery in 18 tertiary hospitals across 10 provinces in China. Patients receiving volatile anaesthetics received at least one volatile anaesthetic (sevoflurane, isoflurane, desflurane), and those who received non-volatile anaesthetics did not receive any volatile anaesthetic. Binary logistic regression analyses were conducted, and propensity score-matching (PSM) and subgroup analyses were also applied.

ELIGIBILITY:
Inclusion Criteria:

Geriatric surgical patients ≥65 years old Non-selective cardiac surgery Non-neurosurgical

Exclusion Criteria:

1. underwent reoperation within 7 days
2. ASA classification of Ⅳ or above
3. history of serious mental illness or long-term use of psychotropic drugs
4. patients either died or were transferred to the intensive care unit within 7 days of the surgery
5. subjects with missing covariate data

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (aged ≥ 65 years) who completed the anxiety and depression assessment on the seventh day after the elective noncardiac, non-neurosurgical surgery were included in this study.
Sampling Method: Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Depression | Depression within 7 days of surgery
  Primary outcomes were depression Patient Health Questionnaire 9 (PHQ-9).The PHQ-9 is a nine-item questionnaire for screening on the presence of depressive symptoms and monitoring depression severity. Items were scored on a four-point scale with total scores ranging from zero to twenty-seven. Scores were defined as: ≥5 mild, ≥10 moderate, and ≥15 severe level of depression. The recommended screening cutoff was ≥10, corresponding with at least a moderate level of depression. The higher the score, the worse the situation. The total score ranges from 0 to 27, and higher scores indicate more depressive symptoms.

SECONDARY OUTCOMES:
Anxiety | Anxiety within 7 days of surgery
  The GAD-7 is a seven-item questionnaire for screening on the presence of generalized anxiety disorder and assessing its severity. Items were scored on a four-point scale with total scores ranging from zero to twenty-one. Scores were defined as: ≥5 mild, ≥10 moderate, and ≥15 severe anxiety. The recommended screening cutoff was ≥10, corresponding with at least a moderate level of anxiety. Higher scores mean more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: WEIDONG MI, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided